CLINICAL TRIAL: NCT01912703
Title: The Long-term Neurodevelopmental Outcome After Intraventricular Hemorrhage (IVH)-Grades I-II in Preterm Infants at Ages 1-7 Years
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-297-13
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Premature Infants
MeSH Terms: conditions — Premature Birth | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm infants with IVH Grades I-II: Preterm infants (post-menstrual age 24-35 weeks) who were diagnosed with IVH Grades 1-2 in the neonatal intensive care unit (NICU).
  Interventions: Other: Telephone interview
- Control Group: Preterm infants (post-menstrual age 24-35 weeks) who had no imaging evidence of IVH in the neonatal intensive care unit (NICU).
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — Subjects with incomplete data will be asked to complete a telephone interview

SUMMARY:
It is well-known that preterm delivery can be accompanied by complications. One of these complications is Intraventricular Hemorrhage (IVH). There are four degrees of IVH, according to severity. It is known that IVH Grades 3-4 can cause severe neurodevelopmental outcomes, including cerebral palsy (CP), hemiplegia, lower motor and cognitive skills and social difficulties. It is not known whether IVH Grades I-II have any of these effects and the aim of this study is to determine whether they do have any neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants born at 35 weeks or less
* Underwent at least 1 brain ultrasound
* Diagnosed with IVH Grades 1-2
* Had no other severe illness in NICU
* Had neurodevelopmental follow-up

Exclusion Criteria:

* All others

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born in 2007-2011 at the Hillel Yaffe Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
General Neurodevelopmental Assessment | Seven years
  Retrospective study of preterm infants born in the years 2007-2011 and suffered IVH Grades 1-2 who have undergone a general neurodevelopmental assessment in the Institute for Child Development in Hillel Yaffe Medical Center at ages 1-7. This assessment will indicate whether IVH Grades 1-2 has any neurodevelopmental effect on these children.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel